CLINICAL TRIAL: NCT04401839
Title: Amr Maneuver for Prevention of Postpartum Hemorrhage After Vaginal Delivery in Term Women
Brief Title: Amr Maneuver for Prevention of Postpartum Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 59
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 153 patients received Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby according to the WHO recommendation for both groups in prevention of postpartum haemorrhage,followed by active management of the third stage of labor by administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
  Interventions: Drug: Oxytocin IV shot; Drug: Oxytocin IV drip
- Study group (Active Comparator): 156 patients received Oxytocin 10 IU I.V shot at the time of delivery of the of the anterior shoulder of the baby according to the WHO recommendation .Then oxytocin is stopped and cervical traction (Amr maneuver )is applied.
  Interventions: Drug: Oxytocin IV shot; Procedure: Amr maneuver

INTERVENTIONS:
Drug: Oxytocin IV shot — Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby
Drug: Oxytocin IV drip — administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation
  Arms: Control group
Procedure: Amr maneuver — sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds
  Arms: Study group

SUMMARY:
The patients were divided randomly in to 2 GROUPS:

* control group: 153 patients received Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby according to the WHO recommendation for both groups in prevention of postpartum haemorrhage,followed by active management of the third stage of labor by administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
* study group:156 patients received Oxytocin 10 IU I.V shot at the time of delivery of the of the anterior shoulder of the baby according to the WHO recommendation .Then oxytocin is stopped and cervical traction (Amr maneuver )is applied.

DETAILED DESCRIPTION:
The patients were divided randomly in to 2 GROUPS:

* control group: 153 patients received Oxytocin 10 IU I.V shot administered at the time of delivery of the anterior shoulder of the baby according to the WHO recommendation for both groups in prevention of postpartum haemorrhage,followed by active management of the third stage of labor by administration of oxytocin 5 IU units IM (WHO GDG recommendations,2012) and waiting for signs of placental separation then controlled cord traction (CCT)to the umbilical cord while applying simultaneous counter-pressure to the uterus, through the abdomen(Brandt Andrews maneuver)
* study group:156 patients received Oxytocin 10 IU I.V shot at the time of delivery of the of the anterior shoulder of the baby according to the WHO recommendation .Then oxytocin is stopped and cervical traction (Amr maneuver )is applied.

In the maneuver,sustained traction downward and posteriorly was applied to anterior and posterior lips of the cervix using ovum forceps for approximately 90 seconds. The traction should be adequate to allow the cervix to reach the vaginal introitus. Meanwhile (CCT ) is avoided and watchful waiting for signs of placental separartion till 90 seconds end. Massage is not employed but the fundus is frequently palpaple to insure it doesnot become atonic and filled with blood from placenta separation. In cases whom placental separation did not occur within the 90 seconds, we removed the ovum forceps and waited for 30 min for the placental separation .

ELIGIBILITY:
Inclusion Criteria:

* women who candidate for vaginal delivery at casualty department singleton fetus full term pregnancy ( gestational age of more than 37 weeks).

Exclusion Criteria:

* fetal macrosomia, any case with bleeding tendency e.g: haemorrhagic diseases cases with risk of postpartum haemorrhage as: Peripartun hemorrhage ( placenta previa or placental abruption), anemia or hypertension.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 306 (Estimated)
Dates: Start 2020-05-31 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
postpartum hemorrhage | 24 hours after delivery
  blood loss more than 500 cc after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No